CLINICAL TRIAL: NCT04575350
Title: Intérêt de la réinterprétation Des CNV de Signification Inconnue Mis en évidence Par ACPA
Brief Title: Reinterpretation of CNV With Unknown Significance: a 5-year Retrospective Analysis
Acronym: ReAC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laetitia LAMBERT, Dr, Central Hospital, Nancy, France
Other Study IDs: ReAC
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Genetic Disease; CNV; Genetic Counseling; Array CGH
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: no intervention.
  Interventions: Genetic: reinterpretation of CNV

INTERVENTIONS:
Genetic: reinterpretation of CNV — Reinterpretation of CNV of unknown significance

SUMMARY:
We aim to assess the usefulness of systematic reinterpretation of CNV of unknown significance. To investigate this question we will study all CNV of unknown significance detected between 2010 and 2017.

DETAILED DESCRIPTION:
Array-CGH is a front-line technique in many genetic indications in both prenatal and postnatal settings. It allows the detection of chromosomal rearrangements (duplication or deletion for example) in routine. The interpretation and classification of these copy number variations or CNVs is essential but complex. It requires a systematic and methodical analysis of the variation in the context of the scientific literature. When these revisions do not meet either pathogenicity or benignity criteria, they are referred to as variation of unknown significance (or VUS). They account for a significant proportion of the revisions up to 75% (Palmer et al., 2013).

The detection of VUS does not, in most cases, allow for a diagnosis and often requires the use of other, costly techniques. The human impact may also be significant in the absence of possible genetic counselling (e.g. in the context of a future pregnancy). Reanalysis of an VUS is of major interest for at least two reasons : (1) the first, if it is classified as benign, makes it possible to close the investigation of the variant, to consider other leads without ulterior motives, and to reassure the patient about the absence of pathogenicity of the variant. (2) if the VUS is ultimately pathogenic, this makes it possible to name the disease for the patient, to specify genetic counselling, to avoid further long and costly investigation and possibly to propose treatment.

Currently, VUS can be reanalysed by the laboratory at the request of the prescribing physician or possibly another physician. However, no systematic reanalysis procedure is currently in place.

Although these variations of unknown meanings are frequent and represent an important issue, to our knowledge, no systematic database study has been carried out. Some similar work has nevertheless been carried out over a shorter period or on an ad hoc basis, showing an interest in this type of approach (Palmer et al., 2014).

Indeed, it seems essential to determine the interest of reanalysing such variations in several modes: diagnostic, economic and human.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent for array-CGH (authorization for the conservation of a biological sample and its subsequent use to continue investigations);
* array-CGHcarried out at the genetics laboratory in Nancy between 1st January 2010 and 31th December 2017 (considering the date of validation of the report);
* Identification of variations of unknown clinical significance.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Define the overall rate and per year of reclassification of CNVs after systematic analysis of all those identified as VUS between 2010 and 2016. | between july 2019 and november 2019
  The proportion of pathogenic variants will correspond to the percentage of pathogenic variants among all reclassified variants.

SECONDARY OUTCOMES:
Among the reclassified CNVs, define the proportion of pathogenic variants ; | between july 2019 and november 2019
  The proportion of pathogenic variants will correspond to the percentage of pathogenic variants among all reclassified variants.
Among the CNVs reclassified as pathogens, define the proportion of new diagnoses ; | between july 2019 and november 2019
  The proportion of new diagnoses corresponds to the proportion of patients for whom the pathogenicity is related to the pathology among all resolved pathogenic variants.
Compare the rate of reclassification of CNVs by type (deletion/duplication) | between july 2019 and november 2019
  The type of reclassification is defined either by deletion or by chromosomal duplication
Compare the size of the CNV according to the type of reclassification of the variant. | between july 2019 and november 2019
  in bp
Compare the reclassification rate by type of disease. | between july 2019 and november 2019
  The following types of conditions will be considered: prenatal/postnatal; intellectual disability or neurodevelopmental disorder/malformation/other.

CONTACTS AND LOCATIONS:
Overall Officials: Lambert Laëtitia, MD, PhD, Principal Investigator — CHRU Nancy, Lorraine University
Locations (1):
- Lorraine University, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palmer E, Speirs H, Taylor PJ, Mullan G, Turner G, Einfeld S, Tonge B, Mowat D. Changing interpretation of chromosomal microarray over time in a community cohort with intellectual disability. Am J Med Genet A. 2014 Feb;164A(2):377-85. doi: 10.1002/ajmg.a.36279. Epub 2013 Dec 5. PMID 24311194
- [Derived] Ravel JM, Renaud M, Muller J, Becker A, Renard E, Remen T, Lefort G, Dexheimer M, Jonveaux P, Leheup B, Bonnet C, Lambert L. Clinical utility of periodic reinterpretation of CNVs of uncertain significance: an 8-year retrospective study. Genome Med. 2023 May 23;15(1):39. doi: 10.1186/s13073-023-01191-6. PMID 37221613